CLINICAL TRIAL: NCT00884507
Title: A Dose-ranging, Randomized, Double-blind , Placebo-controlled Study of the Effect of RO5313534, Used as add-on Therapy to Donepezil, on Cognitive Function in Patients With Mild to Moderate Symptoms of Alzheimer's Disease
Brief Title: A Study of RO5313534 as Add-on to Donepezil Treatment in Patients With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WN22018; 2008-004012-13
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- RO5313534 15mg (Experimental)
  Interventions: Drug: RO5313534
- RO5313534 1mg (Experimental)
  Interventions: Drug: RO5313534
- RO5313534 5mg (Experimental)
  Interventions: Drug: RO5313534

INTERVENTIONS:
Drug: Placebo — po daily for 24 weeks
  Arms: Placebo
Drug: RO5313534 — 1mg po daily for 24 weeks
  Arms: RO5313534 1mg
Drug: RO5313534 — 5mg po daily for 24 weeks
  Arms: RO5313534 5mg
Drug: RO5313534 — 15mg po daily for 24 weeks
  Arms: RO5313534 15mg

SUMMARY:
This 4 arm study will assess the efficacy and safety of RO5313534 (MEM3454) versus placebo added to donepezil, in patients with mild to moderate Alzheimer's disease. Following a screening period, patients will be randomized to one of 4 treatments (placebo, or RO5313534 1mg, 5mg or 15mg po daily) with background therapy of donepezil (5mg or 10mg).The anticipated time on study treatment is 6 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/=50 years of age;
* probable Alzheimer's disease;
* MMSE score at screening of 13-22;
* under stable donepezil treatment given at a fixed dose of 5 or 10mg daily for >=4 months prior to baseline;
* not requiring nursing home care, but looked after by a caregiver/carer.

Exclusion Criteria:

* dementia due to condition other than Alzheimer's disease;
* other significant neurological disorder;
* untreated/non-stabilized major depressive disorder;
* bipolar disorder, schizophrenia, or any other serious psychiatric condition.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2009-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-Cog) score | Week 24

SECONDARY OUTCOMES:
CANTAB tests, MMSE total score, ADCS CGIC, Behave-AD-FW, ADCS-ADL, Zarit Burden interview | At intervals up to week 24, then at week 28
AEs, lab parameters, suicidal risk, concomitant medications, physical and neurological examinations. | At intervals to week 24, then at week 28

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (61):
- United States (14):
  - Orange, California
  - Torrance, California
  - Norwalk, Connecticut
  - Delray Beach, Florida
  - Fort Myers, Florida
  - Maitland, Florida
  - Tampa, Florida
  - Paducah, Kentucky
  - Kalamazoo, Michigan
  - Creve Coeur, Missouri
  - Eatontown, New Jersey
  - Albuquerque, New Mexico
  - White Plains, New York
  - Portland, Oregon
- Argentina (2):
  - Buenos Aires
  - Caba
- Australia (3):
  - Hornsby, New South Wales
  - Chermside, Queensland
  - Woodville, South Australia
- Canada (10):
  - Medicine Hat, Alberta
  - Vancouver, British Columbia
  - Kingston, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Peterborough, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Verdun, Quebec
  - Regina, Saskatchewan
- France (4):
  - Montpellier
  - Nice
  - Saint-Herblain
  - Toulouse
- Germany (4):
  - Günzburg
  - Leipzig
  - München
  - Nuremberg
- Italy (3):
  - Napoli, Campania
  - Castellanza, Lombardy
  - Milan, Lombardy
- Mexico (4):
  - Aguascalientes
  - Guadalajara
  - Monterrey
  - Saltillo
- Poland (4):
  - Gdansk
  - Leszno
  - Torun
  - Warsaw
- Bucharest, Romania
- Slovakia (2):
  - Bratislava
  - Michalovce
- Spain (6):
  - Barcelona, Barcelona
  - BArcelon, Barcelona
  - Salt, Girona
  - Madrid, Madrid
  - Málaga, Malaga
  - Barakaldo, Vizcaya
- United Kingdom (4):
  - Blackpool
  - Bradford
  - Glasgow
  - Southampton